CLINICAL TRIAL: NCT04061941
Title: A Prospective Study to Evaluate the Change in Cognitive Function in Stimulant Users
Brief Title: Change in Cognitive Function in Stimulant Users
Acronym: SToP-S_CogFx
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Beat Drugs Fund Association (Unknown)
Responsible Party: Principal Investigator, Dr. Albert Kar-Kin Chung, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: BDF180058
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Dysfunction; Stimulant Use; Methamphetamine Abuse; Cocaine Use; Substance Use
MeSH Terms: conditions — Cognitive Dysfunction; Substance-Related Disorders | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stimulant Users: Stimulant users that fulfill SCID-5 clinician version definition for assessment on stimulant use disorder under DSM-5
  Interventions: Behavioral: Cognitive Assessment

INTERVENTIONS:
Behavioral: Cognitive Assessment — Assessment on cognitive dysfunction using standardised cognitive tests

SUMMARY:
In Hong Kong, methamphetamine use is common and cocaine use has increased steadily over the past few years. While the use of ketamine decreased from 35.8% in 2015 to 13.9% in 2017, methamphetamine and cocaine have become the most commonly used psychotropic substances and account for more than 50% of drug abuses cases in 2017. Among all stimulants, methamphetamine is most commonly used because it releases three times more dopamine than cocaine and the effects can last from eight to twelve hours, compared to two hours for cocaine. On top of its extreme effects, methamphetamine is relatively inexpensive, making it even more accessible to the young population.

Misuse of methamphetamine has long been associated with profound psychological and cognitive disturbance. In reviewing the cognitive data from reasonably well-matched groups of chronic methamphetamine users and healthy controls, the majority of studies have found that chronic methamphetamine users had lower scores on at least some cognitive tests, although some studies are exceptions with entirely nonsignificant differences. A meta-analysis of 17 cross-sectional studies found that chronic methamphetamine users demonstrated significantly lower cognitive scores than healthy controls. The effects were largest for measures of learning, executive functions, memory, and processing speed, although the majority of cognitive domains significantly differed between the groups.

Concerns has been emerging regarding the methodology of the aforementioned results. In particular, the appropriateness of using healthy controls to examine the cognitive effects of stimulant use has been questioned. Much of the published research has fallen victim to using controls with significant baseline differences from the chronic stimulant users, such as years of education. In addition, none of the studies available provided scatter plots of their cognitive data to evaluate the overlap in performance between chronic stimulant users and healthy controls. In fact, many chronic stimulant users have normal cognitive function when compared with normative data. Therefore, the use of the term 'impairment' or 'deficit' in many studies is not fully justified. Another limitation is that it cannot differentiate cognitive weaknesses that may predate stimulant use from those that result from it. Notably, longitudinal studies have shown that childhood deficits in executive function can predict drug abuse in adolescence, suggesting that at least some of the cognitive weaknesses pre-exist in chronic stimulant user. These and other limitations provoked a conclusion that the evidence for cognitive deficits in chronic stimulant users is weak.

In order to overcome the methodological issues observed in previous cross-sectional studies, we propose to conduct a prospective studies to determine the change in cognitive function among stimulant users over time.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 65 years old at the time of enrolment
* Able to read and communicate in English and/or Chinese
* Able to give informed consent
* Using stimulants as the primary psychoactive substance of abuse
* "Repeated" and "Active" stimulant users as defined by Structured Clinical Interview for DSM-5 Disorders (SCID-5)

Exclusion Criteria:

* Age <18 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Had been diagnosed with other Substance Use or Related Disorders with severity ≥4 according to DSM-5, or other psychoactive substance dependence syndrome according to International Classification of Disease (ICD-10)
* Currently taking regular prescribed psychiatric medications, including antipsychotics, antidepressants, mood stabilizers, anti-epileptics, benzodiazepines, hypnotics, and anti-cholinergic medications.
* Had been diagnosed with other DSM-5 disorders including:

  * Neurodevelopmental Disorders
  * Schizophrenia Spectrum and Other Psychotic Disorders
  * Bipolar and Related Disorders
  * Depressive Disorders, Anxiety Disorders, and Obsessive-Compulsive and Related Disorders
  * Dissociative Disorders, Somatic Symptoms and Related Disorders
  * Feeding and Eating Disorders
  * Sleep-wake Disorders
  * Neurocognitive Disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: stimulant users who have been taking stimulants regularly
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-10-21 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment | 12 months
  Measure the change in global cognitive function
Frontal Assessment Battery | 12 months
  Measure the change in executive function
Diagnostic and Statistical Manual of mental disorders 5th edition (DSM-5 )severity of stimulant use disorder | 12 months
  To determine different severity of stimulant use

SECONDARY OUTCOMES:
Frequency of stimulant use | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No